CLINICAL TRIAL: NCT00604877
Title: Effects of Exercise on Endothelial Function in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Frederick M. Ivey, PhD, Assistant Professor, University of Maryland School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0092; 5K01AG019242 (NIH)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Stroke; Cerebrovascular Disorders
Keywords: exercise; glucose metabolism; insulin sensitivity; Vascular Function
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Treadmill Exercise
- 2 (Active Comparator)
  Interventions: Behavioral: Stretching/ROM

INTERVENTIONS:
Behavioral: Treadmill Exercise — 3 times per week for 6 months, with target of 45 minutes at 60-70% heart rate range
  Arms: 1
Behavioral: Stretching/ROM — 3 times per week for 6 months, passive and active stretching and range of motion (ROM) exercises for the upper and lower extremities
  Arms: 2

SUMMARY:
This study examines the hypothesis that 6 months of treadmill aerobic exercise training improves fibrinolysis (clot defense mechanism) and vasomotor function in chronic hemiparetic (muscular weakness or partial paralysis restricted to one side of the body) stroke patients compared to a control intervention, and that these changes are associated with reduced plasma insulin levels and improved insulin sensitivity / glucose metabolism in this population.

DETAILED DESCRIPTION:
Stroke is the leading cause of disability and third leading cause of death in the United States. Each year approximately 750,000 individuals suffer a stroke, after which they remain at high risk for recurrent stroke and cardiovascular events. Incidence of stroke nearly doubles with each successive decade in older adults, with about 90% of strokes occurring in individuals over 55 years of age.

Following stroke, physical inactivity in advancing age increases the incidence of elevated insulin levels and the insulin resistance syndrome, which are powerful factors that heighten risk for recurrent stroke and myocardial infarction (MI) by impairing fibrinolysis and vasomotor reactivity. Currently, prevention of recurrent stroke and MI depends on best medical management, including antiplatelet therapy, which has limited efficacy. Though aerobic exercise training (AEX) has been shown to improve insulin-glucose metabolism, fibrinolysis profiles, and vasomotor reactivity in healthy elderly and type 2 diabetics, there are no data on the effects of AEX on insulin sensitivity and related vascular endothelial cell function in the chronic hemiparetic stroke population. This trial addresses a significant public health gap, in that aerobic exercise rehabilitation therapy has never been systematically studied as a means to improve cardiovascular health profiles in this population.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic Stroke greater than 6 months prior in men or women ages 40-85
* Residual hemiparetic gait deficits
* Already completed all conventional inpatient and outpatient physical therapy
* Adequate language and neurocognitive function to participate in exercise testing and training

Exclusion Criteria:

* Already performing greater than 20 minutes aerobic exercise 3 times per week
* All insulin dependent diabetics; non-insulin dependent diabetics with fasting glucose greater than 180 mg/dl
* Alcohol consumption greater than 2oz. liquor or equivalent per day
* Cardiac history of: (a) unstable angina, (b) recent (less than 3 months) myocardial infarction, (c) symptomatic congestive heart failure, (d) hemodynamically significant valvular dysfunction
* Medical History of: (a) recent (less than 3 months) hospitalization for severe medical disease, (b) PAOD (Peripheral Arterial Obstructive Disease) with claudication, (c) orthopedic or chronic pain condition restricting exercise, (d) pulmonary or renal failure, (e) active cancer, (f) poorly controlled hypertension (greater than 160/100) (g) Anemia defined by hematocrit less than 30
* Neurological History of: (a) dementia with Mini-Mental Status Score less than 23 (less than 17 if education level at or below 8th grade), and diagnostic confirmation by neurologist or geropsychiatrist, (b) severe receptive or global aphasia which confounds testing and training, operationally defined as unable to follow 2 point commands, (c) hemiparetic gait from prior stroke preceding the index stroke defining eligibility, (d) non-stroke neurological disorder restricting exercise (e.g. Parkinson's Syndrome), (e) untreated major depression
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-08; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Resting and Post-Stressor Fibrinolysis | Baseline and 6 months
Cerebral and lower extremity vasomotor reactivity | Baseline and 6 months
Nitric oxide biomarkers | Baseline and 6 months
Fasting insulin, HOMA-IR, post-load insulin response, glucose tolerance, insulin sensitivity, insulin signaling | Baseline and 6 months

SECONDARY OUTCOMES:
Peak aerobic capacity | Baseline and 6 months
Mobility Function (Timed walks etc..) | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Ivey, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Baltimore VA Medical Center/ University of Maryland School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ivey FM, Ryan AS, Hafer-Macko CE, Goldberg AP, Macko RF. Treadmill aerobic training improves glucose tolerance and indices of insulin sensitivity in disabled stroke survivors: a preliminary report. Stroke. 2007 Oct;38(10):2752-8. doi: 10.1161/STROKEAHA.107.490391. Epub 2007 Aug 16. PMID 17702957
- [Background] Ivey FM, Ryan AS, Hafer-Macko CE, Garrity BM, Sorkin JD, Goldberg AP, Macko RF. High prevalence of abnormal glucose metabolism and poor sensitivity of fasting plasma glucose in the chronic phase of stroke. Cerebrovasc Dis. 2006;22(5-6):368-71. doi: 10.1159/000094853. Epub 2006 Aug 3. PMID 16888377
- [Background] Ivey FM, Macko RF, Ryan AS, Hafer-Macko CE. Cardiovascular health and fitness after stroke. Top Stroke Rehabil. 2005 Winter;12(1):1-16. doi: 10.1310/GEEU-YRUY-VJ72-LEAR. PMID 15735997
- [Background] Ivey FM, Gardner AW, Dobrovolny CL, Macko RF. Unilateral impairment of leg blood flow in chronic stroke patients. Cerebrovasc Dis. 2004;18(4):283-9. doi: 10.1159/000080353. Epub 2004 Aug 24. PMID 15331874